CLINICAL TRIAL: NCT04078217
Title: Novel Tools for the Delivery and Assessment of Exercise Programs Adapted to Individuals With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Université du Québec a Montréal (Other)
Collaborators: Weston Brain Institute (Other)
Responsible Party: Principal Investigator, Christian Duval, Professor, Université du Québec a Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CER VN 18-19-38
Record Dates: First submitted 2019-08-15; First posted 2019-09-04 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease
Keywords: home-based exercise program; gait; mobility
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Masking Description: One of the investigator (the research assistant) will not know the type of intervention (technology or booklet), until the last week of testing when the investigator takes back the equipment for intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jintronix (Experimental): Jintronix Rehabilitation System uses Microsoft Kinect cameras to track patient's movements in 3D during exercises. They are programmed as games that are visualized on a TV and for which performance feedback is provided to the participant. Individualized asynchronous supervised home-base exercise program using the Jintronix System, 3 times/week for 12 weeks (36 sessions). A trained kinesiologist will install the system and supervise the exercise program, in person and remotely.
  Interventions: Device: Jintronix
- Control (Active Comparator): Participants in this group will follow an individualized non-supervised home-based exercise program (booklet format). The exercise program will include 3 sessions per week for 12 consecutive weeks, as for Jintronix group. Actually, all movements of the booklet program are selected to match the exercise-games of the technology (similar movement, muscles engagement, etc.). A trained kinesiologist will explain and supervise the exercise program for the first sessions. The communication frequence will be the same as the Jintronix group.
  Interventions: Other: Booklet

INTERVENTIONS:
Device: Jintronix — Participants will perform an exercise program at home through a telerehabilitation platform called Jintronix.
  Arms: Jintronix
Other: Booklet — Home-based exercise program using a paper booklet (not the technology).
  Arms: Control

SUMMARY:
The study will aim to determine whether a technology-based personalized home exercise program delivered asynchronously and supervised remotely by a kinesiologist is more effective in improving gait than a similar home-based exercise program without technology nor remote supervision. The main hypothesis is that the proposed intervention with the technology will provide significant improvements in gait performance and higher adherence/satisfaction over the non-supervised exercise program.

Both groups will be composed of people with Parkinson's disease. They will have the same evaluation pre and post intervention, the same number of visits from the kinesiologist to deliver the exercise program at home. The difference is the information gathered from the technology; for example, the completion level of each training, success or failure of selected exercises, connection to exercise session, etc. In addition, kinesiologist can remotely adjust difficulty of exercise and take action quickly if the participant hasn't logged in the training system.

Total duration for a participant is 16 weeks: pre-evaluation at home and at lab, 12 weeks home-based exercise program, post-evaluation at home and lab (same as before exercise program).

Pre- and post-evaluation: 7 days wearing an Apple watch to measure mobility in participant environment (participant is met at home and continues normal activities), than comes to lab to undergo physical and balance tests, and scans to analyse body composition (fat, muscle and bone structures). Participant needs to be in "off" state when arriving at the lab; not have taken the morning PD medication. Will take it at the lab with breakfast, after the first tests.

DETAILED DESCRIPTION:
The specific aims of this project are: a) to determine whether a technology-based personalized home exercise program delivered asynchronously and supervised remotely by a kinesiologist is more effective in improving gait than a traditional home-based exercise program, b) to assess the system acceptability and satisfaction, c) to examine and compare the impact of both approaches on several secondary outcome measures related to mobility, PD symptom, and quality of life. This study is a prospective randomized controlled single-blinded clinical trial of efficacy of a technology asynchronous assisted supervised tele-exercise program compared to an a traditional home-based exercise program with a booklet.

Interventions:

Control group (CONT): The participants (n=21) included in control group will follow a non-supervised home-based exercise program (booklet format). The exercise program will include 3 physical activity sessions per week for 12 consecutive weeks. This exercise regimen has been shown to be adequate to improve functional capacities in elderly and feasible. Each exercise session will last 40-45 minutes and includes: 1) 5 minutes of warm-up exercises; 2) 15-18 minutes of mobility and balance exercises (e.g. high knees, lateral launches, side steps); 3) 15-18 minutes of strengthening and coordination exercises (e.g. weight transfer and squats, leg extension and balance, lateral shifting, horizontal flexion and extension) and; 4) 5 minutes for cool down/stretching. This exercise protocol was developed based on general guidelines for the prescription of exercises to older adults and, validated in a previous study. The exercise booklet will be introduced and supervised for the first sessions by a trained kinesiologist. Follow-ups by phone will happen at sessions 6, 12 and 18. During these follow-up calls, if the answers are "yes" to the 3 following questions (1. Did the participant perform during the last weeks all the exercise sessions? 2. Did the participant feel safe when performing exercises? 3. Did the participant find easier to perform the exercises compared to the last contact?), then the participant will be invited, but not obligated, to increase the level of difficulty using the option indicated in the booklet.

JIN Group (n=21): The JIN group (n=21) will receive an individualized asynchronous supervised home-base exercise program using the Jintronix System, 3 times/week for 12 weeks (36 sessions). This exercise regimen has shown to be adequate to improve functional capacities in elderly. Briefly, the Jintronix Rehabilitation System (JRS) uses Microsoft Kinect cameras to track patient's movements in 3D during exercises. They are programmed as games that are visualized on a television and for which performance feedback is provided to the participant. Developed by Jintronix system designers in partnership with researchers, the system provides an interactive exergame environment to execute, specialized exercises through specific instructions and real-time feedback. The Jintronix system which includes a computer, the software and a motion capture device will be installed at participants' homes on their own television. A trained kinesiologist will install the system and supervise the exercise program. Participants will be trained to use the system with help of the kinesiologist during the visits. Each exercise session will last 40-45 minutes and includes: 1) 5 minutes of warm-up exercises; 2) 15-18 minutes of mobility and balance exercises (e.g. high knees, lateral launches, side steps); 3) 15-18 minutes of strengthening and coordination exercises (e.g. weight transfer and squats, leg extension and balance, lateral shifting, horizontal flexion and extension) and; 4) 5 minutes for cool down/stretching. Based on the Web-portal daily reports on the performance of the exercise program, the kinesiologist will do online adjustment of the degree of difficulty of the individualized exercises by increasing the number of repetitions, number of series, intensity and range of motion and provide feedback to the participant. This will ensure individualized adaptations and progress throughout the 12-week intervention.

The JIN group will use the Jintronix rehabilitation software to exercise at home whereas the CONT group will use an exercise booklet. Both groups will be free to exercise on the 3 days and times that best suit their schedule, with a mandatory minimum of one day off between sessions. In addition, to counteract human interaction bias, both exercise groups will have the same number and type of contact. The first weeks following the baseline evaluation, 3 to 4 in-person home visits are required to ensure proper and safe execution of exercise protocol (both groups) and the capacity to use the technology (JIN group only). In addition to these visits, 3 follow-up phone calls will be given to allow the kinesiologist to ensure safety and adherence. An emergency contact number will be given to participants for any questions regarding the exercise regimen during the 12-week intervention.

Study workflow and monitoring: After a phone screening to ensure eligibility and obtaining an oral consent to participate, participants will follow 2 baseline visits: 1 at their home and 1 at the "Université du Québec à Montréal" (UQAM). Before the home visit, subjects will be randomized into control (CONT) or Jintronix® (JIN). During the first visit at home, participants will sign an informed consent form. Afterward, the visit will be divided in 2 parts. The first part will serve to complete validated questionnaires (Parkinson's Disease Questionnaire, Short Falls Efficacy Scale-International and Life Space Assessment). The second part is to install the wearable equipment for mobility assessment (Apple watch® and location beacons). Participants will wear the sensor for at least 7 consecutive days. Afterwards, participants will return wearable sensors and location beacons at the UQAM visit. They will arrive in the morning in "off" state (abstinence of medication 12h before appointment) to undergo the motor evaluation, which is the 6-minute walk test, and the Short Physical Performance Battery test. After these, participants will take their medication with a breakfast at the lab. While waiting to be "on" state, investigators will perform the body composition (DEXA) and muscle composition scans (Ct-scan). When the medication is fully in effect, functional capacity and 6-min walk tests will be re-assessed. This will provide us comparison measures. All evaluations will be repeated at the end of the exercise intervention using the same sequence.

Power analysis:

Sample size: Primary outcome measure is the average gait speed assessed during a 6-minute walk test. Based on previous studies, obtaining clinically significant improvement in gait speed needs to show a gain of 0.2m/sec after intervention. Data using the proposed technology yielded significant improvement (JIN:+0,2±0,12m/s vs CONT:0,05 ±0,09m/s; p=0.025). Thus, obtaining a power of 0.80, an alpha of 0.05, with an effect size of 0.5 (which is significantly smaller that the investigators previously obtained (1.37)), this project would need a total sample size of 28 participants (14 per group) to detect clinically significant differences in gait speed changes between two groups. However, considering an attrition rate of 20% (3 out of 14 in each group) and to improve chances to achieve adequate power for secondary outcomes, a sample of 21 participants per group (n=42) will be used. Even if adequate power is not achieved for the secondary outcomes' measures, sample sizes between 24 and 50 are sufficient to calculate the standard deviation of outcome measures gathered during a feasibility study, to estimate the sample size required for hypothesis testing in a randomized control trial (RCT). Thus, calculations will ensure a sufficient power analysis for the primary outcome measure and position the investigators to establish the variability on secondary measures for a larger RCT.

Statistical analyses: Descriptive statistics (means, standard deviations, ranges, normality, and proportions) will be determined for all study variables. The primary outcome, gait speed, will be assessed using a two-way mixed model analysis of variance (ANOVA) where group is the between factor and time is the within factor. Tukey post hoc or Friedman test will be used based on data characteristics. Categorical variables related to the outcome measures (i.e. clinical scales and diary) will be analyzed using χ2 or Fisher exact tests for baseline comparisons. The change in each outcome variable (before and after training) will be modeled in an unadjusted 1-factor (group) analysis of variance, to investigate the effect of interventions. Wearable sensor data will be averaged over multiple days and compared using a two-way mixed model ANOVA as described above, similar to other secondary outcome measures (i.e. DEXA, CT-Scan, etc.). Tukey post hoc or Friedman test will be used based on data characteristics. To examine changes in variability, standard deviations will be averaged over multiple days and compared using the same approach. Finally, exploratory analyses will be performed to examine 1) if the JIN intervention allows to improve on/off periods, 2) the possible effect of age, sex or medication dose on exercise adaptations.

Innovation: Patients with PD are likely to experience a decrease in their daily physical activity (PA) because of physical impairments, fatigue, and apathy. PA is a complement to pharmacological interventions to manage the inherent decline in function associated with the disease. It is well known that PA interventions induce positive effects on physical capacities and more specifically on gait, mobility, posture and balance. However, engaging older adults in PA through different modalities of exercise programs to obtain these benefits is a challenge, as more than half of older adults are inactive physically and patients with PD are even more than older adults. Supervised exercise programs are needed to motivate and engage patients with PD in becoming more physically active in structured and safe ways. Providing access to supervised exercise programs for patients is difficult as they have mobility constrains and they rely on others for their travel. Home Exercise Programs (HEPs) offer potential benefits but are often lacking close supervision and interaction with a healthcare professional. The use of a supervised in-home PA program driven and supported by an exergame such as Jintronix© has the potential to be more impactful and meaningful to patients than traditional HEPs. It can be used independently by them in their own home and do not require the presence of a professional to perform physical activity training. This allows patients to perform exercise as they wish (schedule, day, on/off period etc.) which overall will increase their adherence to the PA program and promote self-engagement and self-management of their PD. The technology provides a unique way to engage patients in PA while ensuring supervision and communication with a health care professional. The proposed works will also innovate by using an ecological mobility measurement approach based on wearable sensors to capture gait and activity metrics under real life conditions for multiples days and link this to medication use. The combination of sensors used (inertial sensor at the ankle, and interior and exterior location sensors) and their packaging into highly usable and wearable form factors is highly innovative and unique. The proposed instrumentation for the measurement approach offers a lot of potential to study the impacts of pharmacological and non-pharmacological interventions on real life functions and activities of patients. It could be of interest to other parties involved in clinical trials on interventions for PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD from a neurologist based on the clinical diagnostic criteria for PD based on the recent work of Postuma and colleagues
* Hoehn and Yahr stages 1 to 3
* lives on the island of Montreal

Exclusion Criteria:

* Unstable medical/psychiatric comorbidities
* History of other movement disorders
* Orthopedic conditions restricting exercise
* Already performing more than 20 minutes of aerobic exercise more than 3 times per week (to avoid prior training effect)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Gait parameters | 6 min walk test
  Distance walked in 6 min (in meters)
Technology feasibility | 12 weeks
  Automated logs from Jintronix system (performance on each exercise-game)
Technology acceptability | 12 weeks
  Automated logs from Jintronix system (compliance)

SECONDARY OUTCOMES:
Ecological activity | Minimum 7 days
  Data from Apple watch & location beacons: (active time and sedentary time)
Ecological mobility | Minimum 7 days
  Data from Apple watch (distance and mode of travel outside of the home)
Functional capacity | 10 minutes
  Short physical performance battery (SPPB): combines results of gait speed, chair stand and balance tests.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Duval, PhD, Principal Investigator — Université du Québec a Montréal
Locations (1):
- Centre de recherche de l'Institut universitaire de gériatrie de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No